CLINICAL TRIAL: NCT02774720
Title: How do we Get People With MCI and Dementia to be Physically Active?
Brief Title: Centre- Versus Home-based Exercise for MCI and Early Dementia
Acronym: CHIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20687
Record Dates: First submitted 2016-04-07; First posted 2016-05-17 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2018-09

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Centre-based physical activity (Experimental): People with Mild Cognitive Impairment (MCI) and early dementia will receive centre-based physical activity for one hour each week for three months, plus at-home prescribed exercise.
  Interventions: Behavioral: Centre-based exercise
- Home-based exercise (Experimental): People with Mild Cognitive Impairment (MCI) and early dementia be prescribed at-home prescribed exercise and will received monthly support phone calls.
  Interventions: Behavioral: Home-based exercise

INTERVENTIONS:
Behavioral: Centre-based exercise — Participants will come to a centre (University of Waterloo or Toronto Rehabilitation Institute) for a one-hour, small group exercise class each week. The classes will include progressive aerobic and resistance exercise. They will be prescribed additional exercise to be performed independently (either at home or in the community).
  Arms: Centre-based physical activity
Behavioral: Home-based exercise — Participants will be prescribed aerobic and resistance exercise to be performed independently (either at home or in the community). They will receive monthly phone calls to discuss achievements and barriers and to tje adjust exercise prescription.
  Arms: Home-based exercise

SUMMARY:
The study is a proof-of-concept, double-blinded randomized, parallel group trial to compare the effectiveness of centre-based and home-based physical activity in helping people with MCI and early dementia meet physical activity recommendations. The primary outcome is achievement of physical activity recommendations. Secondary outcomes include cost-effectiveness and improvements in health and function.

DETAILED DESCRIPTION:
The aim of this trial is to compare the effectiveness of center-based versus home-based physical activity delivery among people with MCI and early dementia and to understand the influence of person and setting characteristics.

OBJECTIVES:

Primary: To compare the effectiveness of centre-based versus home-based physical activity delivery among people with MCI or early dementia, as measured by percent achievement of physical activity guidelines.

Secondary:

(i) To determine the influence of person- and setting-specific factors. (ii) To estimate the cost-effectiveness of centre-based and home-based physical activity.

Exploratory:

i) To compare the effect of centre- and home-based physical activity on other outcomes.

ii) To explore whether participants consider certain aspects of the program to be important to program effectiveness.

METHODS:

The investigators will conduct a 3-month proof-of-concept, double-blinded randomized, parallel group trial to compare the effectiveness of centre-based and home-based physical activity in helping people with MCI and early dementia meet physical activity recommendations.

Participants will be randomized to one of two physical activity delivery options.The goal of both arms will be to have participants reach physical activity guidelines by the end of the 3-month intervention.

Participants who are randomized to centre-based physical activity will attend physical activity programming at a centre (University of Waterloo or Toronto Rehabilitation Institute) once per week for one hour. Additional physical activity will be prescribed at home.

Participants who are randomized to the home-based physical activity will received a physical activity prescription to be completed at home. They will also receive monthly support calls to assess achievements and barriers and to adjust the prescription.

All assessors will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCI or mild dementia
* Mini-Mental State Examination (MMSE)>=23 or Montreal Cognitive Assessment (MoCA)>=18
* 50 years or older
* Stable pharmaceutical regimen >=2 months
* Be able to travel to centre
* Have a care partner or significant other to support home-based exercise
* Ability to walk >=2 minutes
* Adequate English to understand exercise training
* Adequate hearing and vision for cognitive tests
* Able to comply with assessment and training schedule
* Be screened safe for exercise by a physician or certified exercise physiologist

Exclusion Criteria:

* Current moderate or high intensity exercise >=3 times per week
* Unstable cardiovascular disease that precludes exercise
* Musculoskeletal impairments that limit ability to walk
* Pain or other co-morbidities that would limit exercise
* Behavioural issues that would limit exercise training

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Achievement of Physical Activity | 3 months
  Percent achievement of physical activity recommendations (150min/wk of moderate or high intensity physical activity) as objectively measured using an activity monitor.
Change in physical activity | baseline to 3 months
  Change in physical activity as objectively measured using an activity monitor.

SECONDARY OUTCOMES:
Cost-effectiveness | 3 months
  Cost of resource utilization per minute change in physical activity.

OTHER OUTCOMES:
Change in cognitive function as characterized by Alzheimer's Disease Assessment Scale - Cognition (ADAS-Cog) | baseline to 3 months
  Change in continuous scores
Change in cognitive function as characterized by the Stroop task | baseline to 3 months
  Change in continuous scores
Change in cognitive function as characterized by the Trail making task | baseline to 3 months
  Change in continuous scores
Change in cognitive function as characterized by the semantic fluency | baseline to 3 months
  Change in continuous scores
Change in physical function as characterized by the Short Physical Performance Battery (SPPB) scores | baseline to 3 months
  Change in continuous scores
Change in quality of life as measured with the EuroQol five dimensions questionnaire (EQ-5D) | baseline to 3 months
  Change in continuous scores
Change in mood as measured with the Neuropsychiatric Inventory Questionnaire (NPI-Q) (depression/dysphoria, anxiety, apathy/indifference scales) | baseline to 3 months
  Change in scores, number meeting screening criteria for depression
Change in daily function as characterized using the 6-item Disability Assessment for Dementia (DAD-6) | baseline to 3 months
  Change in score
Change in body mass index (BMI) | baseline to 3 months
  Change in score
Change in waist circumference | baseline to 3 months
  Change in score
Change in blood pressure | baseline to 3 months
  Change in number with high blood pressure (>140 systolic blood pressure (SBP), >90 diastolic blood pressure (DBP))

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Research Institute, Toronto, Ontario
  - University of Waterloo, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Middleton LE, Black SE, Herrmann N, Oh PI, Regan K, Lanctot KL. Centre- versus home-based exercise among people with mci and mild dementia: study protocol for a randomized parallel-group trial. BMC Geriatr. 2018 Jan 25;18(1):27. doi: 10.1186/s12877-017-0684-0. PMID 29370756